CLINICAL TRIAL: NCT04488302
Title: A Retrospective Study on Use of Ultrasonography and Cone-Beam Computed Tomography for Evaluating Peri-implant Tissue
Brief Title: Ultrasonography and Cone-Beam Computed Tomography for Peri-implant Tissue Evaluation
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Clinical Associate Professor, University of Michigan
Other Study IDs: HUM00179671
Record Dates: First submitted 2020-07-15; First posted 2020-07-27 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Implant group: Patients with 1 or more implants with CBCT, ultrasound and open-bone images

SUMMARY:
Objectives: Although cone-beam computed tomography (CBCT) is becoming a standard of care in implant therapy, concerns have been raised recently about its limitation in imaging peri-implant tissues due to artifacts. The aim of present study was to demonstrate the complementary role of ultrasound (US), for a comprehensive examination of peri-implant tissues in live humans. Material and Methods: Patients with > 1 implant, a CBCT scan, an US scan, and clinical photographs taken during the open-bone surgery were included. The crestal bone thickness (CBT) and facial bone level (FBL) were measured on both modalities, and direct FBL measurements were also made on clinical images. The correlation plots were made to evaluate the measurement agreements between the 3 methods.

ELIGIBILITY:
Inclusion Criteria:

* the patients had to have ≥ 1 implant with a CBCT scan, US scan, and clinical photographs taken during the surgery, e.g. a revision/explantation surgery due to peri-implantitis or a 2nd stage uncover surgery.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: See eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Crestal bone thickness | up to 100 months after implant surgery.
  facial bone thickness measured at 1 mm apical to bone crest

SECONDARY OUTCOMES:
Facial bone height | up to 100 months after implant surgery.
  facial bone height measured from implant platform

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No share with others